CLINICAL TRIAL: NCT01458054
Title: Phase 1, Open Label Study to Evaluate the Effect of Omeprazole and Ritonavir on GSK2336805 Pharmacokinetics in Healthy Adults
Brief Title: Effect of Omeprazole and Ritonavir on GSK2336805 Pharmacokinetics in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115711
Record Dates: First submitted 2011-10-06; First posted 2011-10-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
Keywords: pharmacokinetics; omeprazole; ritonavir; healthy subjects; drug interaction
MeSH Terms: conditions — Hepatitis C | interventions — GSK2336805; Omeprazole; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Treatment A (Experimental): GSK2336805 60mg x 1 dose (fasted) [Reference Treatment]
  Interventions: Drug: Cohort 1 (GSK2336805 60mg x 1 dose, Omeprazole 40 mg q24h x 4 days, GSK2336805 60 mg x 1 dose and Omeprazole 40 mg x 1 dose)
- Treatment B (Experimental): Omeprazole 40 mg q24h x 4 days (fed)
  Interventions: Drug: Cohort 1 (GSK2336805 60mg x 1 dose, Omeprazole 40 mg q24h x 4 days, GSK2336805 60 mg x 1 dose and Omeprazole 40 mg x 1 dose)
- Treatment C (Experimental): GSK2336805 60 mg x 1 dose and Omeprazole 40 mg on Day 1 (fasted) [Test Treatment]
  Interventions: Drug: Cohort 1 (GSK2336805 60mg x 1 dose, Omeprazole 40 mg q24h x 4 days, GSK2336805 60 mg x 1 dose and Omeprazole 40 mg x 1 dose)
- Treatment D (Experimental): GSK2336805 30mg x 1 dose (fasted) [Reference Treatment]
  Interventions: Drug: Cohort 2 (GSK2336805 30mg x 1 dose, Ritonavir 100mg q12h x 4 days, and Ritonavir 100mg q12h x 1 dose)
- Treatment E (Experimental): Ritonavir 100mg q12h x 4 days (fed)
  Interventions: Drug: Cohort 2 (GSK2336805 30mg x 1 dose, Ritonavir 100mg q12h x 4 days, and Ritonavir 100mg q12h x 1 dose)
- Treatment F (Experimental): GSK2336805 30 mg x 1 dose (fasted) and ritonavir 100mg q12h on Day 1 (fasted) [Test Treatment]
  Interventions: Drug: Cohort 2 (GSK2336805 30mg x 1 dose, Ritonavir 100mg q12h x 4 days, and Ritonavir 100mg q12h x 1 dose)
- Treatment G (Experimental): Ritonavir 100mg q12h x 1 day
  Interventions: Drug: Cohort 2 (GSK2336805 30mg x 1 dose, Ritonavir 100mg q12h x 4 days, and Ritonavir 100mg q12h x 1 dose)

INTERVENTIONS:
Drug: Cohort 1 (GSK2336805 60mg x 1 dose, Omeprazole 40 mg q24h x 4 days, GSK2336805 60 mg x 1 dose and Omeprazole 40 mg x 1 dose) — GSK2336805 and Omeprazole
  Arms: Treatment A; Treatment B; Treatment C
Drug: Cohort 2 (GSK2336805 30mg x 1 dose, Ritonavir 100mg q12h x 4 days, and Ritonavir 100mg q12h x 1 dose) — GSK2336805 and Ritonavir
  Arms: Treatment D; Treatment E; Treatment F; Treatment G

SUMMARY:
This study is a Phase I open label drug interaction study to evaluate the effect of omeprazole and ritonavir on GSK2336805.

DETAILED DESCRIPTION:
This study is a Phase I open label drug interaction study with two objectives. The first objective of this study (Cohort 1) is to determine if the pharmacokinetics of a single dose of GSK2336805 are affected by co-administration with repeat doses of omeprazole, a proton-pump inhibitor that is commonly used by chronic hepatitis C patients .

The second objective of this study (Cohort 2) is to determine if the pharmacokinetics of a single dose of GSK2336805 are affected by co-administration with repeat doses of ritonavir, a HIV protease inhibitor drug that is a potent inhibitor of CYP 3A4.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin greater than or equal to 1.5x Upper Limit of Normal (ULN) (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with values outside the normal range should always be excluded from enrollment.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, oophorectomy, or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Body weight greater than or equal to 50 kilograms for men and greater than or equal to 45 kilograms for women. Body mass index (BMI) between 18.5-32 inclusive will be allowed (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB less than 450; or QTc less than 480 in subjects with Bundle Branch Block

Exclusion Criteria:

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters within a 56 day period.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject's systolic blood pressure is outside the range of 90-140, or diastolic blood pressure is outside the range of 45-90 or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 beats per minute for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):Heart rate less than 45 and greater than 100 bpm for men and less than 50 and greater than 100 bpm for women. PR interval less than 120 and greater than 220. QRS duration less than 70 and greater than 120. QTc interval greater than 450. Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome). Sinus Pauses greater than 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject. Non-sustained or sustained ventricular tachycardia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

PRIMARY OUTCOMES:
area under the plasma concentration time curve from time zero to the last quantifiable time points | 48 hours
  PK parameter
under the plasma concentration time curve from time zero to infinity | 48 hours
  PK parameter
area under the plasma concentration time curve from time zero to 24 hours | 24 hours
  PK parameter
maximum observed concentration | 48 hours
  PK parameter
time to maximum observed concentration | 48 hours
  PK parameter
concentration at 24 hours post-dose | 24 hours
  PK parameter
last measureable concentration | 48 hours
  PK parameter
time of last measurable concentration | 48 hours
  PK parameter
absorption lag time | 48 hours
  PK parameter
the elimination half-life | 48 hours
  PK parameter
apparent oral clearance | 48 hours
  PK parameter
apparent volume of distribution | 48 hours
  PK parameter

SECONDARY OUTCOMES:
Number of subjects with Adverse Events | 24 hours
  Safety parameter
Number of subjects needing concurrent medications | 24 hours
  Safety parameter
Number of subjects with clinical laboratory tests of clinical significance | 24 hours
  Safety parameter
Number of subjects with electrocardiograms with clinically significant values | 24 hours
  Safety parameter
Number of subjects with vital sign measures of clinical significance | 24 hours
  Safety parameter

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 115711 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115711?search=study&study_ids=115711#rs